CLINICAL TRIAL: NCT02015117
Title: A Phase 1 Study of Trametinib in Combination With Radiation Therapy for Brain Metastases
Brief Title: Trametinib With or Without Whole Brain Radiation Therapy in Treating Patients With Brain Metastases
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-02343; NCI-2013-02343 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); OSU 13197; 2013C0115; 9458 (Other: Ohio State University Comprehensive Cancer Center); 9458 (Other: CTEP); P30CA016058 (NIH); U01CA076576 (NIH); UM1CA186712 (NIH)
Record Dates: First submitted 2013-12-16; First posted 2013-12-19 (Estimated); Last update posted 2025-10-23 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Malignant Neoplasm in the Brain
MeSH Terms: conditions — Brain Neoplasms | interventions — trametinib; omipalisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort A (trametinib, whole-brain radiation therapy) (Experimental): Patients receive trametinib PO QD for 4 weeks. Beginning in week 2, patients undergo whole brain radiation therapy five days a week for 3 weeks. Treatment continues for 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Trametinib; Radiation: Whole-Brain Radiotherapy
- Cohort B (trametinib, surgery) (Experimental): Patients receive trametinib PO QD on days 1-14 followed by surgical resection of the tumor.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Procedure: Therapeutic Conventional Surgery; Drug: Trametinib

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Procedure: Therapeutic Conventional Surgery — Undergo surgical resection of the tumor
  Arms: Cohort B (trametinib, surgery)
Drug: Trametinib — Given PO
  Other Names: GSK 1120212; GSK 212; GSK-1120212; GSK-212; GSK1120212; GSK212; JTP 74057; JTP-74057; JTP74057; MEK Inhibitor GSK1120212
Radiation: Whole-Brain Radiotherapy — Undergo whole-brain radiation therapy
  Other Names: WBRT; whole-brain radiation therapy
  Arms: Cohort A (trametinib, whole-brain radiation therapy)

SUMMARY:
This phase I trial studies the side effects and best dose of trametinib with or without whole brain radiation therapy in treating patients with brain metastases. Trametinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Drugs, such as trametinib, may make tumor cells more sensitive to radiation therapy. Giving trametinib with whole brain radiation therapy may be a better treatment for brain metastases.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To identify the maximally tolerated dose of trametinib to be used in combination with whole brain radiation therapy in patients with brain metastases. (Cohort A) II. To quantify trametinib in resected brain metastatic lesions utilizing high performance liquid chromatography/tandem mass spectrometry (LC/MS/MS) and compare to quantification of adjacent tissues: brain margin, arachnoid, and cerebrospinal fluid (CSF). (Cohort B)

SECONDARY OBJECTIVES:

I. To evaluate the tolerability and feasibility of the combination of trametinib and radiation therapy to brain for brain metastases.

II. To evaluate the objective response rate per Response Evaluation Criteria in Solid Tumors (RECIST) criteria of combination trametinib and radiation therapy.

III. To evaluate the local control rate, as measure from the time of study enrollment until the time of death.

IV. To evaluate the neurologic progression-free survival, as measured from the time of study enrollment until the time of progression within the brain or death.

V. To evaluate overall survival, as measured from the time of study enrollment until the time of death.

TERTIARY OBJECTIVES:

I. To quantify cyclin D1, p27, phosphorylated mitogen-activated protein kinase 1 (pERK)-1/2, phosphorylated v-akt murine thymoma viral oncogene homolog 1 (pAKT), phosphatase and tensin homolog gene (PTEN), phosphorylated mammalian target of rapamycin (pMTOR), phosphorylated ribosomal protein S6 kinase (pS6K), and ribosomal protein S6 (pS6) of resected metastatic brain lesions via quantitative immunohistochemistry (IHC) and compare to the IHC profile of the primary tumor.

OUTLINE: This is a dose-escalation study of trametinib. Patients are assigned to 1 of 2 treatment cohorts.

COHORT A: Patients receive trametinib orally (PO) once daily (QD) for 4 weeks. Beginning in week 2, patients undergo whole brain radiation therapy five days a week for 3 weeks. Treatment continues for 4 weeks in the absence of disease progression or unacceptable toxicity.

COHORT B: Patients receive trametinib PO QD on days 1-14 followed by surgical resection of the tumor.

After completion of study treatment, patients are followed up for 4 weeks, every 2 months for 1 year, every 3 months for 3 years, and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed cancer with measurable or evaluable brain metastases by computed tomography (CT) or magnetic resonance imaging (MRI); MRI is preferred, but a CT scan is acceptable for patients that are unable to have an MRI
* Eastern Cooperative Oncology Group (ECOG) performance status 0 -1
* All prior treatment- related toxicities must be Common Terminology Criteria for Adverse Events (CTCAE) (version 5.0) =< grade 1 (except alopecia) at the time of enrollment
* Absolute neutrophil count >= 1.5 x 10^9/L
* Hemoglobin >= 9 g/dL
* Platelets >= 100 x10^9/L
* Prothrombin time (PT)/international normalized ratio (INR) and partial thromboplastin time (PTT) =< 1.5 x upper limit of normal (ULN) unless using warfarin for therapeutic anti-coagulation
* Albumin >= 2.5 g/dL
* Total bilirubin =< 1.5 x ULN
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x ULN
* Creatinine =< 1.5 ULN or calculated creatinine clearance >= 50 mL/min or 24-hour urine creatinine clearance >= 50 mL/min; calculated by the Cockcroft-Gault formula
* Left ventricular ejection fraction (LVEF) >= 50% by echocardiogram (ECHO) or multigated acquisition scan (MUGA); same method as used at baseline must be use throughout the study, ECHO is the preferred method
* Life expectancy of at least 3 months in the opinion of investigator
* Able to swallow and retain orally administered medication and does not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels
* Ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed
* Women of child-bearing potential (WOCBP) must have a negative pregnancy test within 14 days prior to start of study treatment, and counselled on contraception/abstinence while receiving the study treatment; urine or serum human chorionic gonadotropin (HCG) is an acceptable pregnancy assessment; women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; women of child-bearing potential must have a negative serum or urine pregnancy test within 14 days prior to randomization; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of trametinib administration

Exclusion Criteria:

* Prior radiation therapy to the whole brain (prior stereotactic radiosurgery or fractionated stereotactic radiation therapy to focal areas is allowed)
* Evidence of leptomeningeal metastases
* Urgent need of treatment to prevent acute neurologic deterioration
* Radiosensitive primary tumor such as small cell lung cancer, germ cell tumors, lymphoma, leukemia, or multiple myeloma
* History of another malignancy that makes determination of the source of the brain metastases uncertain
* History of interstitial lung disease or pneumonitis
* Any major surgery, extensive radiotherapy, chemotherapy with delayed toxicity, biologic therapy, or immunotherapy within 14 days prior to enrollment and/or daily or weekly chemotherapy with the potential for delayed toxicity within 14 days prior to enrollment
* Use of other anti-cancer therapies within five half-lives from the previous dose of the prior anti-cancer therapy preceding enrollment and during the study
* Symptomatic or untreated spinal cord compression
* Have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to trametinib, or excipients or to dimethyl sulfoxide (DMSO)
* Current use of a prohibited medication; the following medications or non-drug therapies are prohibited:

  * Other anti-cancer therapy while on study treatment; (note: megestrol [Megace] if used as an appetite stimulant is allowed)
  * Concurrent treatment with bisphosphonates is permitted; however, treatment must be initiated prior to enrollment; prophylactic use of bisphosphonates in patients without bone disease is not permitted, except for the treatment of osteoporosis
  * Concurrent use of all herbal supplements is prohibited during the study (including, but not limited to, St. John's wort, kava, ephedra [ma huang], gingko biloba, dehydroepiandrosterone [DHEA], yohimbe, saw palmetto, or ginseng)
* Drugs that potently inhibit or induce CYP3A4 should be administered with caution; below are a few examples of the agents:

  * Drugs that may increase exposure of trametinib (CYP3A4 inhibitors):

    * Antivirals: amprenavir, atazanavir, fosamprenavir, indinavir, lopinavir, nelfinavir, ritonavir, saquinavir
    * Antibiotics: clarithromycin, erythromycin, telithromycin, troleandomycin
    * Antifungals: fluconazole, itraconazole, ketoconazole, voriconazole
    * Antidepressants: nefazodone
    * Calcium channel blockers: mibefradil, diltiazem, verapamil
    * Miscellaneous: aprepitant
  * Drugs that may decrease exposure of trametinib (CYP3A4 inducers)

    * Antivirals: efavirenz, nevirapine
    * Antibiotic: rifampin
    * Anticonvulsants: carbamazepine, phenobarbital, phenytoin
  * Caution should be exercised when dosing trametinib concurrently with medications with narrow therapeutic windows that are substrates of CYP2C8; below are a few examples of the agents

    * Drug metabolism potentially affected by trametinib resulting in increased exposure of these substrates

      * 3-hydroxy-3-methyl-glutaryl-CoA (HMG CoA)-reductase inhibitors: cerivastatin
      * Thiazolidinediones: rosiglitazone, pioglitazone
      * Miscellaneous: chloroquine, zopiclone, repaglinide
  * As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* History or current evidence/risk of retinal vein occlusion (RVO) or retinal pigment epithelial detachment (RPED):

  * History of RVO or RPED, or predisposing factors to RVO or RPED (e.g., uncontrolled glaucoma or ocular hypertension, uncontrolled systemic disease such as hypertension, diabetes mellitus, or history of hyperviscosity or hypercoagulability syndromes)
  * Visible retinal pathology as assessed by ophthalmic exam that is considered a risk factor for RVO or RPED such as evidence of new optic disc cupping, evidence of new visual field defects, and intraocular pressure > 21 mm Hg
* History or evidence of cardiovascular risk including any of the following:

  * LVEF < lower limit of normal (LLN)
  * A QT interval corrected for heart rate using the Bazett's formula QTcB >= 480 msec
  * History or evidence of current clinically significant uncontrolled arrhythmias (exception: patients with controlled atrial fibrillation for > 30 days prior to registration are eligible)
  * History of acute coronary syndromes (including myocardial infarction and unstable angina), coronary angioplasty, or stenting within 6 months prior to registration
  * History or evidence of current >= class II congestive heart failure as defined by the New York Heart Association (NYHA) functional classification system
  * Treatment-refractory hypertension defined as a blood pressure of systolic > 140 mmHg and/or diastolic > 90 mmHg which cannot be controlled by anti-hypertensive therapy
  * Patients with intra-cardiac defibrillators
  * Known cardiac metastases
* Known hepatitis B virus (HBV), or hepatitis C virus (HCV) infection (with the exception of chronic or cleared HBV and HCV infection, which will be allowed); patients with human immunodeficiency virus (HIV) are not eligible if on anti-retroviral medications
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnancy or breastfeeding (women of childbearing potential should be advised to avoid pregnancy and use effective methods of contraception; men with a female partner of childbearing potential must have either had a prior vasectomy or agree to use effective contraception; if a female patient or a female partner of a patient becomes pregnant while the patient receives trametinib, the potential hazard to the fetus should be explained to the patient and partner (as applicable); radiation therapy is also contraindicated in pregnancy
* Unable to reliably be immobilized for safe administration of whole brain radiation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-04-28 (Actual); Primary Completion 2020-07-10 (Actual); Study Completion 2026-10-08 (Estimated)

PRIMARY OUTCOMES:
Frequency of dose-limiting toxicities (DLT), defined as the maximum dose level of trametinib where at most 1 of 6 patients experience DLT (Cohort A) | Up to 8 weeks
  Frequency of DLTs will be assessed by assessed according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse (CTCAE) version 5.0. DLTs will be summarized by dose level.
Quantification of trametinib in resected brain metastatic lesions utilizing high performance liquid chromatography/tandem mass spectrometry (Cohort B) | Up to day 28
  Trametinib quantification will also be completed in brain margin, arachnoid, and cerebrospinal fluid.

SECONDARY OUTCOMES:
Overall tolerability and toxicity of the regimen, as assessed by adverse events and their grade and attribution for each dose level, graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse (CTCAE) version 5.0 | Up to 8 weeks
  Will summarize observed adverse events and their grade and attribution for each dose level, and patterns reflecting tolerability of the regimen explored through graphical analysis and descriptive summaries. In addition, overall tolerability and toxicity of the regimen will also be evaluated, including reasons for treatment discontinuation as well as the number of patients who successfully complete treatment will be summarized by dose level.
Objective response rate per Response Evaluation Criteria in Solid Tumors | Up to 3 years
  The overall response rate will be assessed as the number of patients who achieve a partial or complete response to therapy divided by the total number of evaluable patients. Assuming that this measure is binomially distributed, the proportion will be estimated and corresponding 95% binomial confidence intervals generated.
Local control rate | Up to 2 years
  Local control rate will be measured from time of study enrollment until the time of progression within the irradiated site.
Neurologic progression-free survival | Time from study entry to the time of progression within the brain or until time of death, assessed up to 2 years
  Described graphically and quantitatively using the methods of Kaplan and Meier.
Overall survival | Time from study entry to the time of death due to any cause, assessed up to 2 years
  Described graphically and quantitatively using the methods of Kaplan and Meier.
Proportion of patients who complete treatment per protocol | Up to 4 weeks
  Assessed as a measure of tolerability.

OTHER OUTCOMES:
Quantification of cyclin D1, p27, pERK-1/2, pAKT, PTEN, pMTOR, pS6K, and pS6 of resected metastatic brain lesions via immunohistochemistry | Up to day 14
  Will be assessed using immunohistochemistry.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua D Palmer, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- [Derived] Palmer JD, Prasad RN, Fabian D, Wei L, Yildiz VO, Tan Y, Grecula J, Welliver M, Williams T, Elder JB, Raval R, Blakaj D, Haglund K, Bazan J, Kendra K, Arnett A, Beyer S, Liebner D, Giglio P, Puduvalli V, Chakravarti A, Wuthrick E. Phase I study of trametinib in combination with whole brain radiation therapy for brain metastases. Radiother Oncol. 2022 May;170:21-26. doi: 10.1016/j.radonc.2022.03.016. Epub 2022 Mar 31. PMID 35367525